CLINICAL TRIAL: NCT02684461
Title: Phase II Trial of Sequential Consolidation With Pembrolizumab Followed by Nab-paclitaxel After Standard First-Line Induction Chemotherapy in Advanced NSCLC
Brief Title: Phase II Trial of Sequential Consolidation With Pembrolizumab Followed by Nab-paclitaxel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1516
Record Dates: First submitted 2016-02-10; First posted 2016-02-18 (Estimated); Results first posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: lung cancer; PD-1 antibody; immune checkpoint blockade
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — pembrolizumab; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A: Sequential Consolidation (Active Comparator): Completion of four cycles of Sequential Consolidation of Pembrolizumab 200mg every 21 days and then four cycles Nab-paclitaxel 100 mg/mg2 on day 1 and day 8 every 21 days
  Interventions: Drug: Pembrolizumab
- Arm B: Sequential Consolidation (Active Comparator): Completion of 4 cycles of Sequential Consolidation of Nab-paclitexel 100 mg/m2 on day 1 and day 8 every 21 days and then Pembrolizumab 200 mg every 21
  Interventions: Drug: Pembrolizumab
- Arm C: Concurrent Consolidation (Active Comparator): Concurrent Consolidation of Nab paclitaxel 100 mg/m2 on day 1 and day 8 plus Pembrolizumab 200 m5 on day 1 every 21 days for four cycles
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Receive Pembrolizumab 200 mg on day 1 every 21 days for four cycles.
  Receive nab-paclitaxel 100 mg/m2 on day 1 and day 8 every 21 days for four cycles.
  Other Names: Keytruda; nab-paclitaxel

SUMMARY:
The purpose of this research study is to test the effectiveness of three treatment arms that are designed to improve survival in patients with non-small cell lung cancer. Eligible subjects could be randomized to four (4) cycles of chemotherapy followed by immunotherapy, or immunotherapy followed by chemotherapy, or four cycles of chemotherapy plus immunotherapy.

DETAILED DESCRIPTION:
This open-label, three-arm, non-comparative randomized phase II study is designed to evaluate three different sequences of double-consolidation with the humanized monoclonal antibody targeted against cell surface receptor programmed cell death-1 (PD-1), pembrolizumab, and nab-paclitaxel in patients with advanced Non small cell lung cancer post induction chemotherapy. While the goal of each arm is to guarantee exposure to each of these two agents to patients who have not progressed post induction chemotherapy, they do so with different sequence. In ARMs A and B, consolidation is sequential, with either pembrolizumab followed by nab-paclitaxel (ARM A), or nab-paclitaxel followed by pembrolizumab (ARM B). In ARM C, consolidation is concurrent, with the two agents administered concurrently. As of July 24, ARMs B and C are closed, and no patients will be enrolled on this study. ARM A remains open to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for this trial
* Be greater than or equal to 18 years of age on day of signing consent
* Eastern Cooperative Oncology Group Performance Status less than or equal to 1
* Histologically or cytologically confirmed confirmed stage IV (metastatic) non small cell lung cancer as defined by American Joint Committee on Cancer (AJCC). Recurrent but not metastatic disease is allowed if deemed incurable.
* Has completed or scheduled to begin 4-6 cycles of platinum based induction chemotherapy that does not include a taxane
* Induction may contain, but is not require to contain bevacizumab or cetuximab.
* Induction with a platinum doublet plus another biologic agent will be allowed following review by the University of North Carolina principal investigator that thee is no additional risk to the subject

NOTE: Evaluable disease is not required for study entry (patients with complete response or response sufficient to preclude measurable lesions are not excluded; such patients will be evaluated for progression free survival and overall survival, but not response)

* Demonstrate adequate organ function (defined in protocol). All screening labs should be performed within 14 days of treatment initiation.
* Recovered from all reversible toxicities related to their previous treatment (other than alopecia) less than or equal to grade 1 or baseline; exceptions to this criteria may be allowed at the discretion of the overall principal investigator for toxicities that are not expected to be exacerbated by pembrolizumab or nab paclitaxel
* Patients with brain metastases may participate if they have undergone appropriate treatment for the lesion)s), are at least two weeks post treatment without evidence for post-treatment progression, have no significant neurologic symptoms, and no longer require steroids for the reason of brain metastases
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for greater than 1 year. The two birth control methods can be two barrier methods or a barrier method plus a hormonal method to prevent pregnancy. Subjects should start using birth control from study Visit 1 throughout the study period up to 120 days after the last dose of study therapy.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Patients with epidermal growth factor receptor (EGFR) mutations expected to be sensitive to epidermal growth factor receptor (EGFR) inhibitors and patients with Echinoderm Microtubule-Associated Protein like 4 anaplastic lymphoma kinase (EML4/ALK) translocations are excluded, unless all available FDA approved targeted therapy options have been utilized. NOTE: In contrast to the above a patient with an EGFR mutation who has been treated with a first-generation and third generation TKIs and then with four cycles of carboplatin plus pemetrexed would be eligible
* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1. Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has had a prior monoclonal antibody within 4 weeks prior to study day 1 or who has not recovered from adverse events due to agents administered more than 4 weeks earlier. Exceptions to these criteria may be allowed at the discretion overall principal for toxicities that are not expected to be exacerbated by pembrolizumab or nab-paclitaxel
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents; subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Has inadequate home environment or social support to safely complete the trial procedures
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-programmed cell death-1 (PD-1) , anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Known hypersensitivity to protein bound paclitaxel
* Has received prior therapy with any taxane chemotherapy
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)
* Has known active Hepatitis B or Hepatitis C
* Has received a live vaccine within 30 days prior to the first dose of trial treatment
* Has a history of non-infectious pneumonitis that required steroids or evidence of interstitial lung disease or current active, non-infectious pneumonitis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared Weiss, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (5):
- United States (5):
  - UNC Lineberger Comprehsive Cancer Center, Chapel Hill, North Carolina
  - Rex Cancer Center, Raleigh, North Carolina
  - Rex Cancer Center of Wakefield, Raleigh, North Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Sequential Consolidation: Completion of four cycles of Sequential Consolidation of Pembrolizumab 200mg every 21 days and then four cycles Nab-paclitaxel 100 mg/mg2 on day 1 and day 8 every 21 days
  Pembrolizumab: Receive Pembrolizumab 200 mg on day 1 every 21 days for four cycles.
  Receive nab-paclitaxel 100 mg/m2 on day 1 and day 8 every 21 days for four cycles.
- Arm B: Sequential Consolidation: Completion of 4 cycles of Sequential Consolidation of Nab-paclitexel 100 mg/m2 on day 1 and day 8 every 21 days and then Pembrolizumab 200 mg every 21
  Pembrolizumab: Receive Pembrolizumab 200 mg on day 1 every 21 days for four cycles.
  Receive nab-paclitaxel 100 mg/m2 on day 1 and day 8 every 21 days for four cycles.
- Arm C: Concurrent Consolidation: Concurrent Consolidation of Nab paclitaxel 100 mg/m2 on day 1 and day 8 plus Pembrolizumab 200 m5 on day 1 every 21 days for four cycles
  Pembrolizumab: Receive Pembrolizumab 200 mg on day 1 every 21 days for four cycles.
  Receive nab-paclitaxel 100 mg/m2 on day 1 and day 8 every 21 days for four cycles.
Period: Overall Study
Arm/Group | Arm A: Sequential Consolidation | Arm B: Sequential Consolidation | Arm C: Concurrent Consolidation
Started | 7 | 7 | 6
Completed | 5 | 5 | 6
Not Completed | 2 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Sequential Consolidation | Arm B: Sequential Consolidation | Arm C: Concurrent Consolidation | Total
Number analyzed (Participants) | 7 | 7 | 6 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 4 | 11
  >=65 years | 3 | 4 | 2 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 3 | 8
  Male | 6 | 3 | 3 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 7 | 5 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 3
  White | 4 | 7 | 6 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as the time from day 1 of treatment to death from any cause. Median overall survival was calculated for each arm.
Time Frame: Up to 60 months
Population: All subjects who received at least one dose of treatment were included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Sequential Consolidation | Arm B: Sequential Consolidation | Arm C: Concurrent Consolidation
Number analyzed (Participants) | 7 | 7 | 6
months | 27.6 [1.7 to NA] — insufficient number of events to calculate upper limit | 12.7 [4.4 to NA] — insufficient number of events to calculate upper limit | NA [NA to NA] — Lack of events to calculate median, upper limit and lower limit

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from first day of treatment until disease progression as defined by the response evaluation criteria in solid tumors (RECIST 1.1) and and Immune Related Response Criteria (irRC), or death from any cause death or progression.
  RECIST 1.1 Progressive Disease (PD): >= 20% increase in the sum of the LD of the target lesions, Stable Disease (SD) Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, Nonprogressive disease (NPD): No measurable disease at the entrance of the study or otherwise non measurable disease will be assessed for progression.
  irRC Progressive Disease (irPD), ≥20% increase in tumor burden and minimum 5 mm absolute increase in compared to nadir; for no new non-target or (irNN) and where irPR or irPD are confirmed by a repeat, consecutive assessment no less than 4 weeks later.
Time Frame: Up to 60 months
Population: All subjects who received at least one dose of treatment were included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Sequential Consolidation | Arm B: Sequential Consolidation | Arm C: Concurrent Consolidation
Number analyzed (Participants) | 7 | 7 | 6
months | 10.1 [1.5 to NA] — insufficient number of events to calculate upper limit | 8.4 [1.2 to 9.0] | 10.2 [5.1 to NA] — insufficient number of events to calculate upper limit

3. Secondary Outcome: Overall Rates of Response (ORR)
Description: ORR is defined as the number of subjects with complete response + partial response based on RECIST 1.1 and irRC criteria.
  RECIST 1.1 Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): >=30% decrease in the sum of the longest diameter (LD) of target lesions.
  irRC Complete Response (irCR): Disappearance of all lesions, no new lesions, lymph nodes < 10 mm in short axis, Partial Response (irPR): ≥30% decrease in the sum of target lesions and non-target lesions are irNN.
Time Frame: 6 months
Population: Subjects received assigned treatment arm were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Sequential Consolidation | Arm B: Sequential Consolidation | Arm C: Concurrent Consolidation
Number analyzed (Participants) | 5 | 7 | 6
Participants
  Complete response | 1 | 0 | 1
  Partial response | 1 | 4 | 2
  Stable disease | 2 | 2 | 3
  Progressive disease | 1 | 1 | 0

4. Secondary Outcome: Rates of Response in Arm A and Arm B
Description: Rates of Response is defined percent tumor size reduction based RECIST1.1 and irRC criteria (the latter if applicable) after each component of therapy in Arm A and Arm B.
Time Frame: 6 months
Population: The subject who is in arm A or Arm B, and received at least 1 dose of study treatment were included.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: Sequential Consolidation: Completion of four cycles of Sequential Consolidation of Pembrolizumab 200mg every 21 days and then four cycles Nab-paclitaxel 100 mg/mg2 on day 1 and day 8 every 21 days
  Pembrolizumab: Receive Pembrolizumab 200 mg on day 1 every 21 days for four cycles.
- Arm B: Sequential Consolidation: Completion of 4 cycles of Sequential Consolidation of Nab-paclitexel 100 mg/m2 on day 1 and day 8 every 21 days and then Pembrolizumab 200 mg every 21
  Pembrolizumab: Receive Pembrolizumab 200 mg on day 1 every 21 days for four cycles.
Arm/Group | Arm A: Sequential Consolidation | Arm B: Sequential Consolidation
Number analyzed (Participants) | 5 | 7
Participants
  Complete Response | 1 | 0
  Partial Response | 1 | 3
  Progressive Disease | 1 | 1
  Stable Disease | 2 | 3

5. Secondary Outcome: Toxicity Profile
Description: The toxicity profile is classified and defined by both provider and the participants reported outcomes.
  Clinician assessed toxicity will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 4.0) Participants assessed toxicity will be classified based on the Patient-Reported Outcome version of the CTCAE (PRO-CTCAE).
  Adverse events occurring in greater than two patients or any grade 3 toxicity were included.
Time Frame: 6 months
Population: All participants received any dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Sequential Consolidation | Arm B: Sequential Consolidation | Arm C: Concurrent Consolidation
Number analyzed (Participants) | 7 | 7 | 6
Participants
  Creatinine Increased: number analyzed (Participants) | 2 | 0 | 0
  Creatinine Increased: Grade 1 | 2 | 0 | 0
  Creatinine Increased: Grade 2 | 0 | 0 | 0
  Creatinine Increased: Grade 3 | 0 | 0 | 0
  Dyspnea: number analyzed (Participants) | 2 | 0 | 0
  Dyspnea: Grade 1 | 1 | 0 | 0
  Dyspnea: Grade 2 | 0 | 0 | 0
  Dyspnea: Grade 3 | 1 | 0 | 0
  Adrenal insufficiency: number analyzed (Participants) | 1 | 0 | 0
  Adrenal insufficiency: Grade 1 | 0 | 0 | 0
  Adrenal insufficiency: Grade 2 | 0 | 0 | 0
  Adrenal insufficiency: Grade 3 | 1 | 0 | 0
  Atrial fibrillation: number analyzed (Participants) | 1 | 0 | 0
  Atrial fibrillation: Grade 1 | 0 | 0 | 0
  Atrial fibrillation: Grade 2 | 0 | 0 | 0
  Atrial fibrillation: Grade 3 | 1 | 0 | 0
  Diarrhea: number analyzed (Participants) | 0 | 3 | 0
  Diarrhea: Grade 1 | 0 | 2 | 0
  Diarrhea: Grade 2 | 0 | 1 | 0
  Diarrhea: Grade 3 | 0 | 0 | 0
  Alopecia: number analyzed (Participants) | 0 | 2 | 2
  Alopecia: Grade 1 | 0 | 2 | 1
  Alopecia: Grade 2 | 0 | 0 | 1
  Alopecia: Grade 3 | 0 | 0 | 0
  Anemia: number analyzed (Participants) | 0 | 2 | 0
  Anemia: Grade 1 | 0 | 1 | 0
  Anemia: Grade 2 | 0 | 1 | 0
  Anemia: Grade 3 | 0 | 0 | 0
  Anorexia: number analyzed (Participants) | 0 | 2 | 0
  Anorexia: Grade 1 | 0 | 2 | 0
  Anorexia: Grade 2 | 0 | 0 | 0
  Anorexia: Grade 3 | 0 | 0 | 0
  Paresthesia: number analyzed (Participants) | 0 | 2 | 0
  Paresthesia: Grade 1 | 0 | 2 | 0
  Paresthesia: Grade 2 | 0 | 0 | 0
  Paresthesia: Grade 3 | 0 | 0 | 0
  Peripheral Sensory Neuropathy: number analyzed (Participants) | 0 | 2 | 0
  Peripheral Sensory Neuropathy: Grade 1 | 0 | 1 | 0
  Peripheral Sensory Neuropathy: Grade 2 | 0 | 1 | 0
  Peripheral Sensory Neuropathy: Grade 3 | 0 | 0 | 0
  White Blood Cell Decreased: number analyzed (Participants) | 0 | 2 | 0
  White Blood Cell Decreased: Grade 1 | 0 | 2 | 0
  White Blood Cell Decreased: Grade 2 | 0 | 0 | 0
  White Blood Cell Decreased: Grade 3 | 0 | 0 | 0
  Alkaline Phosphatase Increased: number analyzed (Participants) | 0 | 1 | 0
  Alkaline Phosphatase Increased: Grade 1 | 0 | 0 | 0
  Alkaline Phosphatase Increased: Grade 2 | 0 | 0 | 0
  Alkaline Phosphatase Increased: Grade 3 | 0 | 1 | 0
  Dehydration: number analyzed (Participants) | 0 | 1 | 0
  Dehydration: Grade 1 | 0 | 0 | 0
  Dehydration: Grade 2 | 0 | 0 | 0
  Dehydration: Grade 3 | 0 | 1 | 0
  Neutrophil count decreased: number analyzed (Participants) | 0 | 1 | 0
  Neutrophil count decreased: Grade 1 | 0 | 0 | 0
  Neutrophil count decreased: Grade 2 | 0 | 0 | 0
  Neutrophil count decreased: Grade 3 | 0 | 1 | 0
  Pain: number analyzed (Participants) | 0 | 0 | 2
  Pain: Grade 1 | 0 | 0 | 2
  Pain: Grade 2 | 0 | 0 | 0
  Pain: Grade 3 | 0 | 0 | 0
  Alanine aminotransferase increased: number analyzed (Participants) | 0 | 0 | 1
  Alanine aminotransferase increased: Grade 1 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 2 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 3 | 0 | 0 | 1
  Hyperglycemia: number analyzed (Participants) | 0 | 0 | 1
  Hyperglycemia: Grade 1 | 0 | 0 | 0
  Hyperglycemia: Grade 2 | 0 | 0 | 0
  Hyperglycemia: Grade 3 | 0 | 0 | 1

6. Secondary Outcome: Quality of Life (QOL) End of Treatment
Description: Changes in QOL score for each subject are defined as the difference between the baseline, and at end of treatment.
  QOL will be evaluated using The Functional Assessment of Cancer Therapy-Lung (FACT-Lung) scale at baseline and the end of treatment. The FACT-L is the FACT-G and a lung cancer-specific (LCS) subscale given at baseline and end of treatment. The FACT-G is a 27-item measure of general QOL assessing function in 4 domains: physical well-being, social-family well-being, emotional well-being, and functional well-being. Items are rated by patients on a Likert scale from 0 to 4. Higher scores represent better QOL.
Time Frame: Baseline to End of Treatment (up to 210 Days)
Population: All participants received any dose of study treatment and responded Functional assessment of Cancer Therapy-Lung questionnaires at the baseline and end of treatment (EOT)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Sequential Consolidation | Arm B: Sequential Consolidation | Arm C: Concurrent Consolidation
Number analyzed (Participants) | 5 | 4 | 5
Participants
  FACT- L Score Increased | 4 | 3 | 4
  FACT- L Score Decreased | 0 | 1 | 0
  FACT- L Score did not Change | 1 | 0 | 1

7. Secondary Outcome: Quality of Life (QOL) 7 Weeks
Description: Changes in QOL score for each subject are defined as the difference between the baseline, and at 7 weeks.
  QOL will be evaluated using The Functional Assessment of Cancer Therapy-Lung (FACT-Lung) scale at baseline and 7 weeks. The FACT-L is the FACT-G and a lung cancer-specific (LCS) subscale given at baseline and at end of treatment. The FACT-G is a 27-item measure of general QOL assessing function in 4 domains: physical well-being, social-family well-being, emotional well-being, and functional well-being. Items are rated by patients on a Likert scale from 0 to 4. Higher scores represent better QOL.
Time Frame: Baseline to 7 weeks (40-50 Days)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Sequential Consolidation | Arm B: Sequential Consolidation | Arm C: Concurrent Consolidation
Number analyzed (Participants) | 4 | 5 | 5
Participants
  FACT- L Score Increased | 3 | 3 | 3
  FACT- L Score Decreased | 1 | 2 | 2
  FACT- L Score did not Change | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events are collected from the first day of the study treatment through 30 days following cessation of treatment (Up to 196 days). Serious AE Collection Time Frame: From the first day of the study treatment through 90 days following cessation of treatment (Up to 256 days).
Description: National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 4.0) used for adverse events grading.
Arm/Group | Arm A: Sequential Consolidation | Arm B: Sequential Consolidation | Arm C: Concurrent Consolidation
All-Cause Mortality (participants affected / at risk) | 1/7 | 1/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/7 | 1/7 | 0/6
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Sequential Consolidation (N=7) | Arm B: Sequential Consolidation (N=7) | Arm C: Concurrent Consolidation (N=6)
Hyponatremia (Metabolism and nutrition disorders) | 1 (7) | 0 (0) | 0 (0)
General disorders and administration site conditions (General disorders) | 0 (0) | 1 (7) | 0 (0) — Death on study
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Sequential Consolidation (N=7) | Arm B: Sequential Consolidation (N=7) | Arm C: Concurrent Consolidation (N=6)
Anemia (Blood and lymphatic system disorders) | 5 | 6 (7) | 3
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 | 2 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 2 | 0
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 3 | 2
Blurred vision (Eye disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 1 | 0
Eye disorders - Other, specify (Eye disorders) | 1 | 0 | 0
Glaucoma (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 3 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 3 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 3 | 3 | 2
Edema limbs (General disorders) | 1 | 3 | 1
Fatigue (General disorders) | 6 | 4 | 4
Fever (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 0
Pain (General disorders) | 3 | 0 | 3
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Allergic reaction (Immune system disorders) | 1 | 0 | 0
Gum infection (Infections and infestations) | 1 | 1 | 0
Papulopustular rash (Infections and infestations) | 0 | 0 | 1
Rhinitis infective (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Intraoperative neurological injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 2
Alkaline phosphatase increased (Investigations) | 1 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 3
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Cholesterol high (Investigations) | 1 | 2 | 0
Creatinine increased (Investigations) | 2 | 0 | 1
Investigations - Other, specify (Investigations) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 3 | 5 | 1
Neutrophil count decreased (Investigations) | 2 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 2
White blood cell decreased (Investigations) | 1 | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 2 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 3 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint range of motion decreased lumbar spine (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Aphonia (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 2 | 0
Paresthesia (Nervous system disorders) | 0 | 2 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 2 | 1
Anxiety (Psychiatric disorders) | 2 | 0 | 1
Depression (Psychiatric disorders) | 2 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 0
Hematuria (Renal and urinary disorders) | 0 | 1 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchopulmonary hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 6 | 3
Thromboembolic event (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/61/NCT02684461/Prot_SAP_000.pdf